CLINICAL TRIAL: NCT01234766
Title: A Multicenter, Open Label, Phase II Study of Bendamustine and Rituximab Followed by 90-yttrium (Y) Ibritumomab Tiuxetan for Untreated Follicular Lymphoma (Fol-BRITe Study)
Brief Title: Bendamustine and Rituximab Followed by 90-yttrium (Y) Ibritumomab Tiuxetan for Untreated Follicular Lymphoma
Acronym: Fol-BRITe
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Cephalon (Industry); Spectrum Pharmaceuticals, Inc (Industry)
Responsible Party: Principal Investigator, Frederick Lansigan, Assistant Professor of Medicine, Dartmouth-Hitchcock Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D1015
Record Dates: First submitted 2010-10-06; First posted 2010-11-04 (Estimated); Results first posted 2018-05-14 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-04

CONDITIONS: Lymphoma, Follicular
MeSH Terms: conditions — Lymphoma, Follicular | interventions — Bendamustine Hydrochloride; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Arm (Experimental): Subjects will receive bendamustine and rituximab, followed by 90-yttrium (Y) Ibritumomab Tiuxetan
  Interventions: Drug: Bendamustine; Drug: Rituximab; Radiation: Y-90 ibritumomab

INTERVENTIONS:
Drug: Bendamustine — 90mg/m2, IV - Days 1 and 2 of every cycle
Drug: Rituximab — 375mg/m2, IV - Cycle 1 only: Day -7 (+1 day) Day 1 of every cycle
  Other Names: Rituxan
Radiation: Y-90 ibritumomab — 0.4mCi/kg, IV - Within 4 hours of rituximab, give over 10 minutes

SUMMARY:
The purpose of the study is to learn about the safety and effectiveness of treating follicular lymphoma with bendamustine and rituximab followed by radioimmunotherapy (RIT) using 90-yttrium (Y) ibritumomab tiuxetan.

The researchers will also test blood and bone marrow for the BCL2 gene-Jh that is a commonly found in people with follicular lymphoma (FL) and look at how the BCL2 gene-Jh responds to the study treatment.

Bendamustine is approved by the United States Food and Drug Administration (FDA) for the treatment of chronic lymphocytic leukemia and indolent B-cell non-Hodgkin's lymphoma (NHL) that has progressed during or within six months of treatment with rituximab or a rituximab-containing treatment regimen. Bendamustine is not approved by the FDA to treat follicular lymphoma.

Rituximab is approved by the FDA for the treatment of relapsed or refractory, low-grade or follicular, CD20-positive B-cell non-Hodgkin's lymphoma.

90-yttrium (Y) ibritumomab tiuxetan is approved by the FDA for the treatment of relapsed or refractory, low-grade or follicular B-cell NHL, including rituximab refractory follicular NHL. It is also approved for the treatment of follicular NHL that is previously untreated with radioimmunotherapy and that achieved a partial or complete response to first-line chemotherapy.

Study participants will will receive bendamustine and rituximab for up to 16 weeks. If participants' cancer responds well to the treatment with bendamustine and rituximab, they will receive up to 12 weeks of radioimmunotherapy (RIT). After the RIT is complete, participants will be asked to return to the clinic every 3 months for a maximum of 10 years for follow-up visits.

DETAILED DESCRIPTION:
STUDY OBJECTIVES

Primary Objective

- To determine the complete response (CR) rate and overall response (OR) rate [CR + partial response (PR) rate] to a regimen of bendamustine and rituximab (B-R), followed by radioimmunotherapy (RIT) with 90-yttrium(Y) ibritumomab tiuxetan in subjects with untreated follicular lymphoma.

Secondary Objectives

* To characterize the safety profile of bendamustine and rituximab followed by 90-yttrium(Y) ibritumomab tiuxetan in subjects with untreated follicular lymphoma
* To determine the CR and OR rate after B-R
* To determine the CR and OR rate after 90-yttrium(Y) ibritumomab tiuxetan specifically the conversions from PR to CR
* To determine the progression-free survival (PFS)
* To determine time to next treatment

Exploratory Objectives

* To determine the molecular response after B-R as determined by qualitative polymerase chain reaction (PCR) of BCL2 from blood and bone marrow examination (required after B-R)
* To determine the molecular response after 90-yttrium(Y) ibritumomab tiuxetan radioimmunotherapy from blood and bone marrow examination (required after RIT)

BACKGROUND

Follicular lymphoma

Non-Hodgkin's lymphomas (NHL) encompass a group of malignancies of lymphocytes that vary in their histologic appearance, aggressiveness and response to therapy.

According to the American Cancer Society, NHL is the 6th most common cancer, with more than 50,000 new cases per year. Follicular lymphoma (FL) is the 2nd most common type of NHL accounting for approximately 20% of newly diagnosed NHL. FL is considered an indolent, but, incurable lymphoma. The goals of therapy are to treat symptomatic advanced stage disease to induce a maximum response with minimal toxicity. The optimal treatment of advanced stage follicular lymphoma (FL) remains to be determined. Combination chemotherapy is the standard frontline treatment option for this disease and the alkylating agent cyclophosphamide has been a common backbone in these combinations. The most common treatments for FL in the United States are rituximab combinations with chemotherapy such as cyclophosphamide, vincristine and prednisone (R-CVP) and cyclophosphamide, doxorubicin, vincristine and prednisone (R-CHOP). The NCCN guidelines also include fludarabine-based regimens, and radioimmunotherapy.

With the addition of immunotherapy (rituximab) to chemotherapy, the overall and complete response rates have improved.1-6 Furthermore, there is suggestive evidence that overall survival may be improved.

Radioimmunotherapy (RIT) is also effective as salvage therapy for indolent lymphoma and transformed lymphoma.7-9 In the first-line setting, RIT following chemotherapy can increase the CR rate and PFS.10-12

Rationale of combining bendamustine and rituximab with consolidation 90-yttrium(Y) ibritumomab tiuxetan

As mentioned above, the combination of bendamustine plus rituximab (B-R) appears to be non-inferior to R-CHOP as first-line treatment of indolent lymphomas including follicular and mantle cell lymphomas, while showing a better tolerability profile such as less alopecia, and potentially less cardiotoxicity, making it a rational choice for first line treatment of FL.17 When given after chemotherapy radioimmunotherapy can convert partial responses to complete responses and can prolong the PFS. The Follicular Lymphoma Ibritumomab tiuxetan (FIT) trial of consolidation Yttrium-90-Ibritumomab tiuxetan versus no additional therapy after first remission in advanced follicular lymphoma showed a prolongation of PFS (36 versus 13 months) in the RIT arm.12 The PFS was prolonged regardless of PR or CR after first-line therapy. The primary treatment included CVP, CHOP, fludarabine-based, and chlorambucil, with the minority of patients receiving rituximab. The results also showed that RIT converted 77% patients from PR to CR/unconfirmed CR (CRu).

An abbreviated course of CHOP-R followed by RIT has shown promise in patients with follicular lymphoma in a phase II trial reported recently.11 Of the 60 patients entering this trial 55 patients completed all protocol therapy. The median follow up was 19.7 months (range, 0.26-35.9 months). For intent-to-treat analysis, the complete response (CR) rate after CHOP-R, as assessed by CT and PET imaging, was 40% and 46%, respectively. After RIT, the CR rate improved, as assessed by CT and PET imaging, to 82% and 89%, respectively.

In this current study, we propose a first-line regimen for untreated FL using bendamustine and rituximab (B-R) (bendamustine 90mg/m2 on days 1 and 2 and Rituximab 375mg/m2 on Day 1 of a 28-day [+2 days] cycle) x 4 cycles followed by RIT; Zevalin (formerly Biogen Idec/Cell Therapeutics, now Spectrum).

The advantage of this treatment is that B-R has a better side effect profile including significantly less alopecia and less infectious complications. Currently bendamustine is not FDA-approved for first-line therapy for follicular lymphoma. 90-yttrium(Y) ibritumomab tiuxetan (Zevalin) radioimmunotherapy is FDA approved for patients with previously untreated follicular non-Hodgkin's Lymphoma (NHL), who achieve a partial or complete response to first-line chemotherapy. Evidence suggests that consolidation with RIT leads to a longer PFS. Since this specific combination has not been utilized in the first-line treatment of FL, it warrants investigation in the current study.

This trial will begin to establish a standard of care for the first-line treatment of follicular lymphoma. We hypothesize that bendamustine plus rituximab followed by RIT will contribute to among the highest CR rates seen in follicular lymphoma with relatively low toxicity. Based on the results of this trial, we would aim to open a larger trial for follicular lymphoma in a cooperative group setting, i.e. CALGB.

Correlative Studies Background

The BCL2 gene-Jh rearrangement is the common abnormality in FL t(14;18). This can be assessed by various PCR techniques.18,19

Patients can be assessed for this molecular abnormality in their bone marrow at baseline and following therapy. For instance in a similar Southwest Oncology Group study of chemotherapy followed by radioimmunotherapy using tositumomab/iodine I-131 tositumomab (Bexxar) for follicular lymphoma, patients were asked to undergo serial bone marrow aspirations at study entry, 4 weeks after the sixth cycle of CHOP (just before tositumomab/iodine I-131 tositumomab), and after tositumomab/iodine I-131 tositumomab for PCR testing.20 The mononuclear cell fraction was isolated from marrow aspirates by Ficoll-Hypaque sedimentation and cryopreserved for subsequent batch analysis using a double nested PCR assay to detect the major breakpoint region and the minor cluster region of the BCL2 gene. Samples were initially analyzed by fragment size using ethidium bromide gel electrophoresis of the PCR product and then transferred to nitrocellulose membranes for confirmation of the identity of the BCL2 translocation by Southern blotting. The adequacy of samples was demonstrated using beta-globin as a positive control housekeeping gene. Patients were considered to have attained a molecular remission if their marrow sample at study entry contained a detectable t(14;18) translocation that became undetectable after protocol treatment.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated, histologically confirmed follicular lymphoma classification grade 1, 2 or 3a
* Ann Arbor stages of II to IV with either symptomatic or bulky disease (>5 cm); or disease progression
* 18 years of age or older
* ECOG PS <2
* Normal organ and marrow function defined as below:

Absolute neutrophil count (ANC) >= 1,000/mm3 Platelet count >=100,000/mm3 Patients with ANC less than 1,000/mm3 and/or platelets below 100,000/mm3 are still eligible for study entry as long as there is >50% bone marrow involvement with lymphoma

* Adequate hepatic function
* Adequate renal function
* Measureable disease with at least one lesion measuring > 2cm in its greatest transverse diameter
* Female subjects of childbearing potential must have a negative pregnancy test (urine or serum b-HCG) at screening and within 1 week prior to the start of treatment with Y-90 ibritumomab tiuxetan
* Voluntary written informed consent must be given before performance of any study-related procedure

Exclusion Criteria:

* Prior chemotherapy, immunotherapy, or monoclonal antibody therapy
* Receiving any other investigational agents
* Primary CNS lymphoma
* Known HIV
* Treatment with therapeutic doses of systemic steroids within 4 weeks of beginning study treatment (cycle 1, day -7); topical use of corticosteroids and systemic replacement of corticosteroids for adrenal insufficiency are allowed
* Malignant pleural, pericardial or peritoneal effusions
* Known history of myelodysplastic syndrome (MDS) or found to have MDS
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would, in the judgment of the investigator, limit compliance with study requirements
* Pregnant or lactating female subjects
* Concurrent active malignancy other than lymphoma or history of invasive malignancy within the past 5 years, except completely excised, non-melanoma skin cancer
* Known Hepatitis B and/or Hepatitis C Infection
* Any other condition, that in the judgment of the investigator places the patient at unacceptable risk if he/she were to participant in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2010-10 (Actual); Primary Completion 2021-01 (Actual); Study Completion 2021-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frederick Lansigan, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (4):
- United States (4):
  - Maine Center for Cancer Medicine, Scarborough, Maine
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Duke University Medical Center, Durham, North Carolina
  - Rhode Island Hospital, Providence, Rhode Island

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Single Arm
Started | 39
Completed | 35
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm
Number analyzed (Participants) | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 28
  >=65 years | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 17
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 39

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Complete Response at 3 Years
Description: The primary endpoint is complete response (CR) rate. Historical complete response (CR) rate has been 35%. This rate will be considered as the null hypothesis.
Time Frame: 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 35
Participants | 30

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the start of treatment until 30 days after the last dose of treatment, approximately 7 months.
Arm/Group | Single Arm
All-Cause Mortality (participants affected / at risk) | 0/39
Serious Adverse Events (participants affected / at risk) | 5/39
Other Adverse Events (participants affected / at risk) | 0/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm (N=39)
Basilar pneumonia (Infections and infestations) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1)
Infusion related reaction (General disorders) | 1 (1)
JC Virus/Progressive Multifocal Leukoencephalopathy (Nervous system disorders) | 1 (1)
Secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Chronic myeloid leukemia

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-06): https://cdn.clinicaltrials.gov/large-docs/66/NCT01234766/Prot_SAP_000.pdf